CLINICAL TRIAL: NCT06845488
Title: Application of Virtual Reality Technology to Treatment of Social Anxiety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Katherine A. Loveland, Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-16-0518
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Autism Spectrum Disorder; Social Anxiety Disorder
Keywords: Virtual reality; psychotherapy
MeSH Terms: conditions — Autism Spectrum Disorder; Phobia, Social

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Virtual Reality (VR) assisted Cognitive Behavior Therapy (CBT) (Experimental)
  Interventions: Behavioral: CBT; Device: VR
- CBT alone (Active Comparator)
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — Participants will receive will receive 12 weeks of weekly CBT for Social Anxiety, including an intervention to improve conversational skills. The CBT for Social Anxiety will include "imaginal exposure", which is a way of using the imagination to work with situations that produce anxiety. Participants will also receive a mindfulness intervention.
Device: VR — The VR software, the Virtual Communicator (VC) consists of a highly realistic avatar that interacts with the client in one of several situations. The therapist controls its gestures, facial expressions, body movements, and speech and builds and saves modular combinations of gestures and facial expressions that can be assembled in any order to create a conversational interaction. The software has two adult avatars of ambiguous race/ethnicity, male and female. The VC is delivered without a headset interactively over the internet, on a secure, password-protected connection that increase access by not requiring headsets and not requiring the client to come to the office. The VC can be done in English, or in Spanish where appropriate. Treatment will be done for 12 sessions. The VR software is used to provide CBT exposures to reduce anxiety and also to practice social interactions.
  Arms: Virtual Reality (VR) assisted Cognitive Behavior Therapy (CBT)

SUMMARY:
The purpose of this study is to compare CBT VR exposure + VR social skills treatment to CBT Imaginal exposure + mindfulness, in reducing the severity of social anxiety in adults with autism and social anxiety (SA), to identify characteristics associated with benefitting from the CBT-VR treatment and to assess acceptability and feasibility of the VR intervention for patients receiving it and use findings to improve methods and to prepare for a community based pragmatic trial.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD) (diagnosed by a qualified professional)
* verbal and literate in English or Spanish
* average or greater intellectual ability, based on history and interview
* able to operate a computer (Windows or Mac).

Exclusion Criteria:

* current or historical severe mental illness such as schizophrenia, bipolar disorder, or severe depression
* intellectual disability or a learning disability that would interfere with participating (e.g., unable to read)
* unable use the technology or do not have access to the technology
* unable to read

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety as assessed by the Liebowitz Social Anxiety Scale (LSAS) | Baseline, 3 weeks, 6 weeks, 9 weeks, 12 weeks, post treatment (about 4 weeks after end of treatment))
  This is a 24 item questionnaire, each is assessed in 2 ways measuring both fear/anxiety and avoidance related to specific social situations, giving a total of 48 ratings across the scale. The questions are scored from 0 (none) to 3 (severe) for a score range of 0-144 higher score indicating worse outcome.
Change in anxiety as assessed by the Social Interaction Anxiety Scale (SIAS) | Baseline, 3 weeks, 6 weeks, 9 weeks, 12 weeks, post treatment (about 4 weeks after end of treatment)
  This is a 20 item questionnaire and each is scored on a likert scale from 0(not at all characteristic of me)-4(Extremely characteristic of me), maximum score of 80,higher score indicating worse outcome
Change in anxiety as assessed by the Social Phobia Scale (SPS) | Baseline, 3 weeks, 6 weeks, 9 weeks, 12 weeks, post treatment (about 4 weeks after end of treatment)
  This is a 20 item questionnaire and each is scored on a likert scale from 0-4, maximum score of 80 , higher score indicating worse outcome
Change in anxiety as assessed by the The Severity Measure for Social Anxiety Disorder (SMSAD) scale | Baseline, 3 weeks, 6 weeks, 9 weeks, 12 weeks, post treatment (about 4 weeks after end of treatment)
  This is a 10 item questionnaire and each is scored from 0(never) to 4(all of the time) for a maximum score of 40, higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Loveland, PhD, Principal Investigator — The University of Texas Health Science Center at Houstom
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No